CLINICAL TRIAL: NCT01043458
Title: A Single Dose Study of the Safety, Tolerability, and Pharmacokinetics of ABT-126 in Stable Subjects With Schizophrenia
Brief Title: Pharmacokinetic Study of ABT-126 in Stable Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Hana Florian, MD / Associate Medical Director, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M11-108
Record Dates: First submitted 2009-10-21; First posted 2010-01-06 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-09

CONDITIONS: Schizophrenia
Keywords: Pharmacokinetics
MeSH Terms: conditions — Schizophrenia | interventions — ABT-126

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): ABT-126 Low Dose
  Interventions: Drug: ABT-126
- 2 (Experimental): ABT-126 High Dose
  Interventions: Drug: ABT-126
- 3 (Experimental): Placebo for ABT-126
  Interventions: Drug: Placebo for ABT-126

INTERVENTIONS:
Drug: ABT-126 — ABT-126 Low Dose & ABT-126 High Dose
  Arms: 1; 2
Drug: Placebo for ABT-126 — Matching Placebo for Arms 1 & 2
  Arms: 3

SUMMARY:
A study to investigate the process by which ABT-126 is absorbed, distributed, metabolized and eliminated by the body of stable schizophrenic volunteers receiving treatment with an atypical antipsychotic.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed informed consent;
* Current diagnosis of schizophrenia;
* Clinically stable on the same single second-generation (atypical) antipsychotic for the past 8 weeks;
* Meets study-specific criteria for Positive and Negative Syndrome Scale (PANSS);
* Females are not pregnant, not breast-feeding;
* Females are post-menopausal or surgically sterile or practicing birth control;
* Males are surgically sterile or agree to be sexually inactive or use barrier method of birth control

Exclusion Criteria:

* Diagnosis of schizoaffective disorder;
* Diagnosis with mental retardation;
* Subject has a substance dependence disorder that has not been in sustained remission for at least 1 year;
* Acute psychosis hospitalization within past 6 months;
* Bipolar disorder, manic episode, dementia, obsessive-compulsive disorder, or drug-induced psychosis or current major depressive disorder;
* Current clozapine treatment;
* Suicidal ideation or behavior;
* BMI of 39 or greater;
* Relevant drug sensitivity or allergy;
* Positive hepatitis or HIV test result; positive urine screen for drugs of abuse or alcohol;
* Recent clinically significant illness/infection or surgery;
* Recent blood product transfusion, donation or loss of 5 mL/kg of blood;

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Duration of study
ABT-126 levels in blood (plasma) | Pre-dose to 144 hours post-dose
Clinical laboratory tests, vital signs and electrocardiogram (ECG) | Pre-dose to 72 hours post-dose

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Site Reference ID/Investigator# 25423, Glendale, California
  - Site Reference ID/Investigator# 24322, San Antonio, Texas